CLINICAL TRIAL: NCT04220320
Title: The Success of Labor Induction Based on a Modified BISHOP Score Compared to Classic BISHOP Score and Cervical Length in Transvaginal Sonography.
Brief Title: The Success of Labor Induction Based on a Modified BISHOP Score.
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal investigator, Rambam Health Care Campus
Other Study IDs: 0622-19-RMB
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Gynecological Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Classic BISHOP score: Gynecological evaluation based on vaginal examination including cervical dilatation, effacement, texture, station and position.
  Interventions: Diagnostic Test: Vaginal examination.
- Modified BISHOP score: Gynecological evaluation based on vaginal examination including cervical dilatation and effacement alone.
  Interventions: Diagnostic Test: Vaginal examination.
- Cervical Length: Gynecological evaluation based on cervical length measured by transvaginal sonography.
  Interventions: Diagnostic Test: Transvaginal sonography.

INTERVENTIONS:
Diagnostic Test: Vaginal examination. — Cervical properties as evaluated by a vaginal examination.
  Groups: Classic BISHOP score; Modified BISHOP score
Diagnostic Test: Transvaginal sonography. — Cervical length as evaluated by a transvaginal sonography.
  Groups: Cervical Length

SUMMARY:
Pregnant women at term will be divided randomly into 3 groups:

1. Gynecological evaluation based on classic BISHOP score.
2. Gynecological evaluation based on a modified BISHOP score.
3. Gynecological evaluation based on cervical length as measured by transvaginal sonography.

After gynecological evaluation, women will undergo induction of labor based on obstetric evaluation according to the group they were part of.

DETAILED DESCRIPTION:
Women presenting to the obstetric emergency room for follow-up for various obstetric/other medical conditions over 37 weeks' gestation that are candidates for labor induction will receive an explanation regarding the study and sign informed consent.

The women will be divided randomly into 3 groups:

1. Gynecological evaluation based on classic BISHOP score.
2. Gynecological evaluation based on a modified BISHOP score.
3. Gynecological evaluation based on cervical length as measured by transvaginal sonography.

After gynecological evaluation, women will undergo induction of labor based on obstetric evaluation according to the group they were part of.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies.
* Candidates for vaginal delivery.

Exclusion Criteria:

* Multiple pregnancies.
* Candidates for cesarean section.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female.
Study Population: Pregnant women over 37 weeks' gestation that are candidates for induction of labor for obstetric/other medical indications.
Sampling Method: Non-Probability Sample
Enrollment: 758 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Time to delivery | Up to 72 hours.
  The time from induction commencement to delivery of the newborn.

SECONDARY OUTCOMES:
BISHOP score after primary induction. | Up to 24 hours.
  BISHOP score after primary induction. BISHOP is not an abbreviation and is just the name of the score. The minimum score is 0 and the maximum score is 13. The higher the score, the more favorable the cervix is considered before induction of labor.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Healthcare Campus
Locations (1):
- Rambam healthcare campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No